CLINICAL TRIAL: NCT02241044
Title: Ivision of Gastroenterology, Department of Internal Medicine, Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan
Brief Title: Argon Plasma Coagulation for Bleeding Peptic Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Huay-Min Wang, Division of Gastroenterology, Department of Internal Medicine, Kaohsiung Veterans General Hospital, Kaohsiung,Taiwan, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS98-CT8-13
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Bleeding Ulcers
Keywords: argon plasma coagulation, bleeding peptic ulcer
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- the Combined group (Active Comparator): The Combined group patients received Argon plasma coagulation therapy, PSD-60/Endoplasma (Olympus Corporation, Tokyo, Japan), following distilled water injection at index endoscopy. Then participants were treated with intravenous pantoprazole (Pantoloc i.v., Nycomed GmbH, Singen, Germany) 40 mg every 12 hours during the first 3 days, followed by oral pantoprazole (Pantoloc, Takeda GmbH, Oranienburg, Germany) 40 mg daily until the end of 56-day study period.
  Interventions: Device: Argon plasma coagulation; Device: Distilled water
- the Injection group (Placebo Comparator): Injection group patients underwent distilled water alone at index endoscopy. Then patients were treated with intravenous pantoprazole (Pantoloc i.v., Nycomed GmbH, Singen, Germany) 40 mg every 12 hours during the first 3 days, followed by oral pantoprazole (Pantoloc, Takeda GmbH, Oranienburg, Germany) 40 mg daily until the end of 56-day study period.
  Interventions: Device: Distilled water

INTERVENTIONS:
Device: Argon plasma coagulation — Argon plasma coagulation therapy was realized by an Olympus electrosurgical unit/APC unit (PSD-60/Endoplasma, Olympus Corporation, Tokyo, Japan), and its catheters were 2.3mm and 3.5 mm equipped with different endoscope channels.7 APC treatment used a coagulation mode at gas flow/power settings of 1.5L/min and 40 watt for duodenal ulcers and 40-60 watt for gastric ulcers.10 Operative distance between the probe and target bleeding ranged from 2 to 8 mm. Air warranted to be sucked frequently at endoscopy in an attempt at decrease of APC-induced smoke and gastric decompensation, with appropriate treatment of high-risk bleeding ulcers.
  Other Names: PSD-60/Endoplasma (Olympus Corporation, Tokyo, Japan)
  Arms: the Combined group
Device: Distilled water — Distilled water was then applied in aliquots of 0.5-2.0 mL, at and around the site of target bleeding, up to 25.0 ml if necessary. Injection amount was determined by endoscopists according to ulcer or vessel size and its location.

SUMMARY:
Background:

A second endoscopic method added to injection therapy is recommended for high-risk bleeding peptic ulcers. Many endoscopic devices have been proved as useful hemostatic instruments, whereas the hemostatic efficacy of argon plasma coagulation (APC) has not been widely investigated.

Aim:

This study was designed to know whether additional APC treatment could influence the hemostatic efficacy after endoscopic injection therapy in treating high-risk bleeding ulcers.

Methods:

From October 2010 to January 2012, eligible patients who had high-risk bleeding ulcers were admitted to our hospital. They prospectively randomly underwent either APC therapy plus distilled water injection or distilled water injection alone. Pantoprazole infusion was conducted during the fasting period after endoscopy and orally for 8 weeks to encourage ulcer healing. Episodes of rebleeding were retreated with endoscopic combination therapy. Patients who did not benefit from retreatment underwent emergency surgery or transarterial embolization (TAE).

DETAILED DESCRIPTION:
Patients and methods Study cohort Patients with acute upper gastrointestinal bleeding (AUGIB) who were admitted to Kaohsiung Veterans General Hospital between January 2011 and January 2012 were screened. Inclusion criteria were (i) over 20 years of age and (ii) patients with high-risk peptic ulcer bleeding. Acute hemorrhage from upper gastrointestine was defined as classical presentation with hematemesis, coffee-ground emesis, and/or melena. High-risk bleeding ulcers were defined as participants with stigmata of a bleeding visible vessels (eg, spurting, oozing), a non-bleeding visible vessels (NBVV) or adherent clot.4 A NBVV at endoscopy was defined as a raised red, red-blue or pale hemispheric vessel protruding from the ulcer bed, without active bleeding. An adherent clot was defined as an overlying blood clot that was resistant to vigorous irrigation.

Exclusion criteria were as follows: (i) the presence of another possible bleeding site (eg, gastroesophageal varix, gastric cancer, reflux esophagitis); (ii) coexistence of actively severe ill diseases (eg, septic shock, stroke, myocardial infarction, surgical abdomen); (iii) treatment with an anticoagulant (eg, warfarin); (iv) pregnancy; (v) the presence of operated stomach or; (vi) refusal to participate in the study.

In current study, baseline characteristics of both study groups were collected at the first 24 hours after admission. Some definitions of events were expressed herein: smoking was defined as inhalation of smoke from burning tobacco daily in recent 3 months; habitual consumption of alcohol was defined as participants imbibing alcohol twice or more per week in recent 3 months; shock was considered systolic blood pressure less than 90 mm Hg or diastolic less than 60 mmHg, and heart rate over 100 beats per minute; comorbid diseases included unresolved malignancy, diabetes mellitus, liver cirrhosis, uremia, congestive heart failure, chronic pulmonary obstructive disease and pneumonia; and coagulopathy was defined as prothrombin time > 14 seconds and/or activated partial thromboplastin time > 45 seconds.

Randomization In this prospective, parallel-group, randomized controlled trial, eligible patients were randomized into two groups using opaque-sealed envelopes numbered according to a table of random numbers before the fist therapeutic endoscopy (index endoscopy): the Combined group and the Injection group. Informed consent was obtained from each enrolled participant. Combined group patients received APC therapy following distilled water injection at index endoscopy. Injection group patients underwent distilled water alone at index endoscopy. Thereafter both treatment groups were treated with intravenous pantoprazole (Pantoloc i.v., Nycomed GmbH, Singen, Germany) 40 mg every 12 hours during the first 3 days, followed by oral pantoprazole (Pantoloc, Takeda GmbH, Oranienburg, Germany) 40 mg daily until the end of 56-day study period. Primary end point was rebleeding. Secondary end points included initial hemostasis, the need for surgery, transfusion requirements, the period of hospitalization, severe adverse event (stricture, obstruction or perforation) and death at 30 days postrandomization.

ELIGIBILITY:
Inclusion Criteria:

* (i) over 20 years of age and (ii) patients with high-risk peptic ulcer bleeding.

Exclusion Criteria:

* (i) the presence of another possible bleeding site (eg, gastroesophageal varix, gastric cancer, reflux esophagitis); (ii) coexistence of actively severe ill diseases (eg, septic shock, stroke, myocardial infarction, surgical abdomen); (iii) treatment with an anticoagulant (eg, warfarin); (iv) pregnancy; (v) the presence of operated stomach or; (vi) refusal to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
rebleeding | up to 30 days
  Rebleeding was observed for a 30-day study period. One or more the following criteria were considered as evidence of recurrent bleeding: aspiration of fresh blood from a nasogastric or orogastric tube; pulse rate over 100 beats per minute; a drop in systolic blood pressure exceeding 30 mmHg; or continue coffee ground emesis or melena with a decline in hemoglobin of at least 2g/dL.

SECONDARY OUTCOMES:
mortality | up to 30 days
  All-cause deaths were recorded.
Surgery | up to 30 days
  the need for surgery wihtin 30 days
sever adverse events | up to 30 days
  Namely, stricture, obstruction and perforation

CONTACTS AND LOCATIONS:
Overall Officials: Huay-Min Wang, MD, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Kaohsiung Veterans General Hospital
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Wang HM, Tsai WL, Yu HC, Chan HH, Chen WC, Lin KH, Tsai TJ, Kao SS, Sun WC, Hsu PI. Improvement of Short-Term Outcomes for High-Risk Bleeding Peptic Ulcers With Addition of Argon Plasma Coagulation Following Endoscopic Injection Therapy: A Randomized Controlled Trial. Medicine (Baltimore). 2015 Aug;94(32):e1343. doi: 10.1097/MD.0000000000001343. PMID 26266385